CLINICAL TRIAL: NCT07108764
Title: Effect of Intraoperative Infusion of Either Lidocaine or Dexmedetomidine on Regional Cerebral Oxygen Saturation and Postoperative Delirium in Elderly Patients Undergoing Abdominal Surgeries
Brief Title: Intraoperative Infusion of Either Lidocaine or Dexmedetomidine on Regional Cerebral Oxygen Saturation and Postoperative Delirium in Elderly Patients Undergoing Abdominal Surgeries
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Dina Hamdy Alhassanin, Assistant Lecturer of Anesthesiology, Surgical Intensive Care and Pain Medicine, Faculty of Medicine, Tanta University, Tanta, Egypt., Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 36265MD399/4/25
Record Dates: First submitted 2025-07-31; First posted 2025-08-07 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-07

CONDITIONS: Intraoperative Infusion; Lidocaine; Dexmedetomidine; Cerebral Oxygen Saturation; Postoperative Delirium; Elderly Patients; Abdominal Surgeries
MeSH Terms: conditions — Emergence Delirium | interventions — Lidocaine; Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lidocaine group (Experimental): Patients will receive an IV bolus (50 ml) of lidocaine (1mg/kg) diluted with saline over 10 min before induction of anesthesia. This will be followed by intraoperative lidocaine infusion in a dose of 1.5mg /kg/hr till the end of surgery.
  Interventions: Drug: Lidocaine
- Dexmedetomidine group (Experimental): Patients will receive an IV bolus (50 ml) of dexmedetomidine in dose 0.5 μg/kg over 10 min before induction of anesthesia. This will be followed by intraoperative dexmedetomidine infusion in a dose of 0.3 μg/kg/hr till the end of surgery.
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Lidocaine — Patients will receive an IV bolus (50 ml) of lidocaine (1mg/kg) diluted with saline over 10 min before induction of anesthesia. This will be followed by intraoperative lidocaine infusion in a dose of 1.5mg /kg/hr till the end of surgery.
  Arms: Lidocaine group
Drug: Dexmedetomidine — Patients will receive an IV bolus (50 ml) of dexmedetomidine in dose 0.5 μg/kg over 10 min before induction of anesthesia. This will be followed by intraoperative dexmedetomidine infusion in a dose of 0.3 μg/kg/hr till the end of surgery.
  Arms: Dexmedetomidine group

SUMMARY:
This study aims to compare the effect of intraoperative infusion of either lidocaine or dexmedetomidine on the incidence of postoperative delirium (POD) in elderly patients undergoing major surgeries. It also aims to evaluate the impact of both medications on intraoperative regional cerebral oxygen saturation (rSO₂).

DETAILED DESCRIPTION:
Postoperative delirium (POD) is a significant complication in elderly patients undergoing major surgery, with an incidence ranging from 10% to 50%, depending on patient and surgical factors.

Regional cerebral oxygen saturation (rSO₂), measured using near-infrared spectroscopy (NIRS), provides a real-time, non-invasive marker of cerebral perfusion. Previous studies have demonstrated that intraoperative declines in rSO₂ are associated with an increased risk of POD.

Lidocaine, an amide local anesthetic, has been shown to reduce neuroinflammation, improve microcirculation, and exert neuroprotective effects. It has been associated with low postoperative pain, reduced opioid consumption, and improved cognitive outcomes.

Dexmedetomidine, an α2-adrenergic agonist, is known for its sedative, analgesic, and sympatholytic effects. It has been shown to enhance cerebral perfusion, improve rSO₂, and reduce POD incidence.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 65years old.
* Both sexes.
* Physical status classification of II - III according to the American Society of Anesthesiologists (ASA).
* Undergo elective non-cardiac surgeries.

Exclusion Criteria:

* History of mental illness, neurological illness, or scoring less than 8 using the abbreviated mental test (AMT) before operation.
* Severe hearing or visual impairment that may interfere with communication.
* Severe renal or hepatic dysfunction.
* Patients on central nervous system (CNS) medications (antipsychotics, anticonvulsants, antiparkinsonian, antidepressants).
* Contraindications to lidocaine or dexmedetomidine [e.g., allergy, severe bradycardia, atrioventricular (AV) block].

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-04-17 (Actual); Primary Completion 2027-04-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of postoperative delirium | Three days after surgery
  Incidence of postoperative delirium (POD) will be recorded.

SECONDARY OUTCOMES:
Regional cerebral oxygen saturation | Till end of surgery (Up to 2 hours)
  Regional cerebral oxygen saturation (rScO2) will be recorded using cerebral oximetry at the baseline, 5 min after induction of general anesthesia, then every 20 min till the end of surgery.
Degree of pain | 24 hours postoperatively
  Postoperative numerical rate scale (NRS) score will be recorded on admission to the post-anesthesia care unit (PACU), at six h, 12h, and 24h postoperatively.
Postoperative opioid consumption | 24 hours postoperatively
  Rescue analgesia in the from 3 mg IV morphine (mg) will be given if the numerical rate scale (NRS) is ≥ 4 repeated with 10 10-minute lock-out interval till the NRS becomes less than 3.
Heart rate | Till end of surgery (Up to 2 hours)
  Heart rate will be recorded at baseline, after induction, after 15 min, then every 15 min till the end of surgery.
Mean arterial blood pressure | Till end of surgery (Up to 2 hours)
  Mean arterial blood pressure will be recorded at baseline, after induction, after 15 min, then every 15 min till the end of surgery.
Incidence of adverse effects | 24 hours postoperatively
  Incidence of adverse effects such as nausea, vomiting, and respiratory depression will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, El-Gharbia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.